CLINICAL TRIAL: NCT02549508
Title: Comparison Study Using APAP With and Without SensAwake in Patients With OSA and PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CIA 134
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnea (OSA); Post-Traumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- AutoCPAP with SensAwake On, then SenAwake Off (Experimental): Participants will start AutoCPAP treatment with SensAwake on for 4 weeks. After 4 weeks, the will cross over to SensAwake off for another 4 weeks.
  Interventions: Device: AutoCPAP with SensAwake On; Device: AutoCPAP with SensAwake Off
- AutoCPAP with SensAwake Off, then SensAwake On (Experimental): Participants will start AutoCPAP treatment with SensAwake Off for 4 weeks. After 4 weeks, the will cross over to SensAwake On for another 4 weeks.
  Interventions: Device: AutoCPAP with SensAwake On; Device: AutoCPAP with SensAwake Off

INTERVENTIONS:
Device: AutoCPAP with SensAwake On — The comfort feature 'SensAwake' will be turned on
Device: AutoCPAP with SensAwake Off — The comfort feature 'SensAwake' will be turned off

SUMMARY:
The purpose of this research is to examine the application of AutoCPAP with and without SensAwake in subjects with OSA and Post-Traumatic Stress Disorder (PTSD), and evaluate whether patients achieve better sleep quality and compliance with SensAwake, compared to the same treatment without SensAwake.

DETAILED DESCRIPTION:
Conceptually, awareness of pressure occurs only during wakefulness. Thus reducing the pressure during wakefulness may improve therapy comfort and potentially adherence without compromising therapy efficacy. SensAwake™ is a unique pressure relief technology developed by Fisher & Paykel Healthcare which detects irregularity in the flow signal indicative of the transition from sleep to wake. When the transition from sleep to wake is detected the device promptly reduces the pressure to help facilitate a return to sleep.

It is hypothesised that AutoCPAP with SensAwake will improve patient comfort and compliance in the PTSD and OSA patients who are naïve to CPAP therapy.

The investigators will not be blinded to the study. The participants will be blinded to the study.

ELIGIBILITY:
Inclusion Criteria:

Male and female subjects > 18 years Diagnosed with OSA by a practicing sleep physician, within the last six months Diagnosed with post-traumatic stress disorder as diagnosed by a behavioral health professional, and quantified by McChord PTSD checklist All races and ethnicities will be included Naïve to CPAP therapy (has not used CPAP within the last 5 years)

Exclusion Criteria:

< 18 years of age if mental status is questionable, the patient will be excluded at the discretion of the consenting provider Unable/unwilling to follow the directions necessary for CPAP use Patients contraindicated for CPAP/AutoCPAP, at the discretion of the consenting provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron B Holley, MD, Principal Investigator — Walter Reed National Military Medical Center; Rebecca Thomson, MA, Study Chair — Fisher & Paykel Healthcare
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holley A, Shaha D, Costan-Toth C, Slowik J, Robertson BD, Williams SG, Terry S, Golden D, Andrada T, Skeete S, Sheikh K, Butler G, Collen JF. A randomized, placebo-controlled trial using a novel PAP delivery platform to treat patients with OSA and comorbid PTSD. Sleep Breath. 2020 Sep;24(3):1001-1009. doi: 10.1007/s11325-019-01936-x. Epub 2019 Nov 6. PMID 31691105

RESULTS

PARTICIPANT FLOW:
Groups:
- AutoCPAP With SensAwake On First, Then SensAwake Off: Randomized participants in this group will experience SensAwake On first while using AutoCPAP for the first 4 weeks of the intervention.
  After 4 weeks, participants will cross over to the opposite arm and complete 4 weeks with SensAwake off while using AutoCPAP.
- AutoCPAP With SensAwake Off First, Then SensAwake On: Randomized participants in this group will experience SensAwake Off first while using AutoCPAP for the first 4 weeks of the intervention.
  After 4 weeks, participants will cross over to the opposite arm and complete 4 weeks with SensAwake on while using AutoCPAP.
Period: Overall Study
Arm/Group | AutoCPAP With SensAwake On First, Then SensAwake Off | AutoCPAP With SensAwake Off First, Then SensAwake On
Started | 47 | 38
Completed | 33 | 21
Not Completed | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- AutoCPAP With SensAwake On First, Then SensAwake Off: Randomized participants in this group will experience SensaAwake On first while using AutoCPAP for the first 4 weeks of the intervention.
  After 4 weeks, participants will cross over to the opposite arm and complete 4 weeks with SensAwake off while using AutoCPAP.
- AutoCPAP With SensAwake Off First, Then SensAwake On: Randomized participants in this group will experience SensaAwake Off first while using AutoCPAP for the first 4 weeks of the intervention.
  After 4 weeks, participants will cross over to the opposite arm and complete 4 weeks with SensAwake On while using AutoCPAP.
- Total: Total of all reporting groups
Arm/Group | AutoCPAP With SensAwake On First, Then SensAwake Off | AutoCPAP With SensAwake Off First, Then SensAwake On | Total
Number analyzed (Participants) | 47 | 38 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.0) | 37.7 (8.6) | 37.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 40 | 33 | 73
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 47 | 38 | 85

OUTCOME MEASURES:

1. Primary Outcome: Adherence (Hours on Therapy)
Description: Hours per night averaged over total time period measured.
Time Frame: 4 weeks
Measure: Mean (Full Range); unit: Hours/night
Groups:
- AutoCPAP With SensAwake On: Analysis of all participants who completed the AutoCPAP with SensAwake on arm.
- AutoCPAP With SensAwake Off First: Analysis of all participants who completed the AutoCPAP with SensAwake off arm
Arm/Group | AutoCPAP With SensAwake On | AutoCPAP With SensAwake Off First
Number analyzed (Participants) | 29 | 25
Hours/night | 1.1 [1.1 to 4.8] | 0.5 [0.0 to 2.7]

2. Secondary Outcome: Sleep Quality (Epworth Sleepiness Scale (ESS)
Description: The ESS is a validated questionnaire that assesses an idnviduals likelihood of falling asleep in a variety of given situations (such as having a conversation with someone or stopped a red light while driving.) Each question is given a rating between 0 and 3, with 0 being no chance of falling asleep and 3 being high chance of falling asleep. Answers are then summed together to determine the level of sleepiness an individual is experiencing with a maximum score of 24. The higher the score, the more sleepy the person is. From a clinical perspective an ESS score of 0-10 indicates a normal level sleepiness, a score of 11-14 indicates mild sleepiness, a score of 15-17 indicates moderate sleepiness and a score of 18+ indicates severe sleepiness. Results below are reported as a mean change from baseline in which negative scores indicate reduction in ESS from baseline (less sleepiness). Positive scores indicate increase in ESS from baseline (more sleepiness.)
Time Frame: Change from Baseline after 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- AutoCPAP With SensAwake Off: Analysis of all participants who completed the AutoCPAP with SensAwake off arm
Arm/Group | AutoCPAP With SensAwake On | AutoCPAP With SensAwake Off
Number analyzed (Participants) | 29 | 25
score on a scale | -2.4 (4.5) | -3.0 (4.4)

3. Secondary Outcome: Insomnia Severity Index (ISI)
Description: ISI; 0-7 = No clinically significant insomnia, 8-14 = Sub threshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe). Results reported in mean change from baseline. Negative scores indicate improvement in ISI, positive scores indicate increase in ISI.
Time Frame: Change from Baseline after 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AutoCPAP With SensAwake On | AutoCPAP With SensAwake Off
Number analyzed (Participants) | 29 | 25
score on a scale | -4.2 (4.5) | -4.4 (4.7)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- AutoCPAP With SensAwake On: Includes data for all participants who were exposed at any point of the 8 week study to SensAwake On. Due to drop outs, not all participants were exposed to this intervention.
- AutoCPAP With SensAwake Off: Includes data for all participants who were exposed at any point of the 8 week study to SensAwake Off. Due to drop outs, not all participants were exposed to this intervention.
Arm/Group | AutoCPAP With SensAwake On | AutoCPAP With SensAwake Off
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72
Other Adverse Events (participants affected / at risk) | 0/71 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT02549508/Prot_SAP_000.pdf